CLINICAL TRIAL: NCT03043989
Title: Two Independent Phase 1b Cohorts of Docetaxel or Cabazitaxel in Combination With the Potent CYP3A4 Inhibitor, Clarithromycin
Brief Title: Cohorts of Docetaxel or Cabazitaxel in Combination With the Potent CYP3A4 Inhibitor, Clarithromycin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Technology Development Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J16144; IRB00117591 (Other: JHM IRB)
Record Dates: First submitted 2017-01-26; First posted 2017-02-06 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: docetaxel; cabazitaxel; phase 1b; castration-resistant; bone metastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; cabazitaxel; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Docetaxel and clarithromycin combination (Active Comparator): Docetaxel will be administered by intravenous infusion over 1 hour every 3 weeks on day 1 of each (3 week) cycle for a total of 18 weeks.
  Clarithromycin will be administered orally at 500mg twice a day for 3 days per cycle on days -1, 1, and 2.
  Interventions: Drug: Docetaxel; Drug: Clarithromycin
- Cabazitaxel and clarithromycin combination (Active Comparator): Cabazitaxel will be administered by intravenous infusion over 1 hour every 3 weeks on day 1 of each (3 week) cycle for a total of 18 weeks.
  Clarithromycin will be administered orally at 500mg twice a day for 3 days per cycle on days -1, 1, and 2.
  Interventions: Drug: Cabazitaxel; Drug: Clarithromycin

INTERVENTIONS:
Drug: Docetaxel — 6 infusions of Docetaxel with 18 doses clarithromycin
  Arms: Docetaxel and clarithromycin combination
Drug: Cabazitaxel — 6 infusions of Cabazitaxel with 18 doses clarithromycin
  Other Names: JEVTANA
  Arms: Cabazitaxel and clarithromycin combination
Drug: Clarithromycin — 18 doses of clarithromycin with either Docetaxel or Cabazitaxel

SUMMARY:
This clinical trial is being conducted to recommend a safe and tolerable phase 2 dose of docetaxel or cabazitaxel when combined with clarithromycin in men who have developed castrate-resistant prostate cancer.

In the castrate-resistant setting, resistance to taxane therapy inevitably develops. Men who develop resistance to taxanes have a very poor prognosis, and few treatment options.

It is believed that CYP enzymes contribute to docetaxel and cabazitaxel resistance in metastatic prostate cancer, and this resistance can be mitigated through pharmacologic CYP inhibition. In this study a potent CYP3A inhibitor, clarithromycin, will be co-administered concurrently with either docetaxel or cabazitaxel, whose systemic metabolism is dependent of CYP3A4, with the intent to overcome resistance to taxanes.

DETAILED DESCRIPTION:
This is a dose-escalation study designed to determine the maximum tolerated dose of docetaxel or cabazitaxel when given in combination with clarithromycin. Eligible patients will be assigned to docetaxel or cabazitaxel, based on which drug they were previously administered prior to study entry. Enrollment to dose levels will be in a 3+3 cohort design until the maximum tolerated dose is achieved.

Docetaxel or cabazitaxel will be administered on day 1 of each (3 week) cycle for a total of 6 cycles. Subjects in both arms will be administered clarithromycin on days -1, 1 and 2 of each 3 week cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Men with metastatic castrate-resistant prostate cancer (prostate cancer progressing despite castrate levels of testosterone <50 ng/dL), using standard measures of progression defined by PCWG2
2. Have received at least 4 cycles of docetaxel or cabazitaxel, and less than ten, with two consecutive rising PSA values, checked at least 7 days apart. No PSA decline in last 42 day
3. Bone disease documented by either: a positive bone scan, CT scan, or MRI; or biopsy-proven bony metastases
4. Age ≥18 years
5. ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
6. Have normal organ and marrow function defined as:

   * absolute neutrophil count ≥1,500/mcL
   * platelets ≥100,000/mcL
   * total bilirubin (within normal institutional limits)
   * AST/ALT ≤ 2.5 × ULN (or ≤ 1.5 x ULN in conjunction with alk phos >2.5 x ULN for Docetaxel
   * AST ≤ 1.5 x ULN for Cabazitaxel
   * creatinine clearance-no minimum for Docetaxel
   * creatinine clearance- ≥ 30 mL/min/1.73 m2 for Cabazitaxel
7. No evidence of clinical progression, in the form of increased lesions on cross-sectional imaging, or new cancer-attributable symptoms or worsening of existing symptoms
8. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients who have residual toxicities > Grade 2 attributed to taxane therapy, except for neuropathy, who are excluded if > grade 1
2. Patients who are receiving any other investigational agents or have within the last 28 day.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to clarithromycin or taxanes
4. Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Received more than 10 cycles of docetaxel [for docetaxel cohort only] or 6 of cabazitaxel [for cabazitaxel cohort only]
7. Last docetaxel or cabazitaxel dose > 6 weeks prior to enrollment
8. Patients with a documented history of QT prolongation or ventricular cardiac arrhythmia, including torsades de pointes, or taking drugs that are known to prolong the QT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 years
Escalate dose up the maximum tolerated dose achieved, and initiate this as the recommended phase 2 dose of docetaxel and of cabazitaxel when it is combined with clarithromycin. | 3 years

SECONDARY OUTCOMES:
Compare docetaxel OR cabazitaxel exposure (maximal [Cmax] when combined with the strong CYP3A4 inhibitor clarithromycin to historic controls. | 3 years
Compare docetaxel OR cabazitaxel exposure ( total [AUC]) when combined with the strong CYP3A4 inhibitor clarithromycin to historic controls. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Carducci, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No